CLINICAL TRIAL: NCT00148954
Title: Rhythm ID Going Head-to-head Trial
Brief Title: RIGHT: Rhythm ID Going Head-to-Head Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR-CA-032105-T; RIGHT
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2011-12-26 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Tachycardia
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Implantable Cardioverter Defibrillator - Boston Scientific (Active Comparator): VITALITY 2 ICD
  Interventions: Device: VITALITY 2 Implantable Cardioverter Defibrillator
- Implantable Cardioverter Defibrillator - Medtronic (Active Comparator): Selected Medtronic family ICD
  Interventions: Device: Medtronic Implantable Cardioverter Defibrillator

INTERVENTIONS:
Device: VITALITY 2 Implantable Cardioverter Defibrillator — VITALITY 2 ICD
  Arms: Implantable Cardioverter Defibrillator - Boston Scientific
Device: Medtronic Implantable Cardioverter Defibrillator — Maximo, Marquis, Intrinsic, Virtuoso, or Entrust ICD
  Arms: Implantable Cardioverter Defibrillator - Medtronic

SUMMARY:
RIGHT is a randomized, prospective, two-arm study that will assess the differential efficacy of VITALITY 2 implantable cardioverter defibrillators (ICDs) using Rhythm ID™ versus selected Medtronic ICDs.

DETAILED DESCRIPTION:
RIGHT will compare the incidence of Ventricular Tachycardia/Fibrillation (VT/VF) therapies delivered for Supraventricular Tachycardia (SVT) episodes using VITALITY 2 devices with Rhythm ID™ to that of ICDs employing other rhythm discrimination algorithms. Appropriateness of therapies will be assessed after independent adjudication of all VT/VF events leading to therapy. Comparisons will be made between device manufacturers across patient populations receiving either a dual- or single-chamber device.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet current indications for an ICD
* Patients who sign and date a Patient Informed Consent form prior to the implant visit
* Patients who remain in the clinical care of the enrolling physician in approved centers
* Patients who are able to tolerate ICD programming as specifically prescribed in the study protocol

Exclusion Criteria:

* Patients who are in third degree heart block
* Patients whose life expectancy is less than 12 months
* Patients who have other cardiac surgeries or procedures planned but not yet performed during the duration of the study
* Patients who are currently enrolled in another investigational study or registry that would directly impact the treatment or outcome of the current study
* Patients who are younger than 18 years of age
* Patients who are mentally incompetent and cannot sign a Patient Informed Consent form or comply with the study
* Patients who are pregnant or plan to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1962 (Actual)
Dates: Start 2005-07; Primary Completion 2009-03 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gold, MD, PhD, Principal Investigator — Medical University of South Carolina; Ron Berger, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Berger RD, Lerew DR, Smith JM, Pulling C, Gold MR. The Rhythm ID Going Head to Head Trial (RIGHT): design of a randomized trial comparing competitive rhythm discrimination algorithms in implantable cardioverter defibrillators. J Cardiovasc Electrophysiol. 2006 Jul;17(7):749-53. doi: 10.1111/j.1540-8167.2006.00463.x. PMID 16836672
- [Derived] Gold MR, Ahmad S, Browne K, Berg KC, Thackeray L, Berger RD. Prospective comparison of discrimination algorithms to prevent inappropriate ICD therapy: primary results of the Rhythm ID Going Head to Head Trial. Heart Rhythm. 2012 Mar;9(3):370-7. doi: 10.1016/j.hrthm.2011.10.004. Epub 2011 Oct 4. PMID 21978966

RESULTS

PARTICIPANT FLOW:
Groups:
- VITALITY 2: VITALITY 2 ICD
- Medtronic Family: Selected Medtronic family devices
Period: Overall Study
Arm/Group | VITALITY 2 | Medtronic Family
Started | 985 | 977
Completed | 678 | 677
Not Completed | 307 | 300

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VITALITY 2 | Medtronic Family | Total
Number analyzed (Participants) | 985 | 977 | 1962
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 489 | 482 | 971
  >=65 years | 496 | 495 | 991
Age Continuous [Mean (Standard Deviation); unit: years] | 64.3 (12.4) | 64.4 (12.0) | 64.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 223 | 197 | 420
  Male | 762 | 780 | 1542
Region of Enrollment [Number; unit: participants]
  United States | 915 | 909 | 1824
  Europe | 65 | 63 | 128
  Canada | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Inappropriate Ventricular Tachycardia (VT)/Ventricular Fibrillation (VF) Therapy (Shock or Antitachycardia Pacing [ATP]) After the Pre-Discharge Visit
Description: An inappropriate therapy is defined as a VT/VF therapy, either shock or antitachycardia pacing (ATP), delivered for a supraventricular tachycardia (SVT). All events for which a VT/VF therapy was delivered and a stored electrogram exists were reviewed by an independent adjudication committee to determine the appropriateness of device rhythm classification and subsequent therapy delivery.
Time Frame: From date of pre-discharge until a minimum of 12 months follow-up until study closure
Measure: Number; unit: Participants
Arm/Group | VITALITY 2 | Medtronic Family
Number analyzed (Participants) | 985 | 977
Participants | 246 | 187
Statistical Analysis 1: Comparison: VITALITY 2 vs Medtronic Family; Test type: Superiority or Other; p = 0.003, Regression, Cox; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [1.11 to 1.62]

2. Secondary Outcome: Time to First Inappropriate Shock Using VITALITY and Selected Medtronic Implantable Cardioverter Defibrillator (ICDs)
Time Frame: Time of event
Reporting Status: Not Posted

3. Secondary Outcome: Positive Predictive Value (PPV) of Ventricular Tachycardia/Fibrillation (VT/VF) Discrimination Algorithms Found in VITALITY 2 and Medtronic Implantable Cardioverter Defibrillators (ICDs)
Time Frame: Time of event
Reporting Status: Not Posted

4. Secondary Outcome: Time to First Inappropriate Therapy for Which the Discrimination Algorithm Found in VITALITY 2 and Medtronic Implantable Cardioverter Defibrillator (ICDs) Inappropriately Classified the Episode
Time Frame: Time of event
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- VITALITY 2; Medtronic Family: This study did not collect serious adverse events
Arm/Group | VITALITY 2 | Medtronic Family
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 535/985 | 508/977
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VITALITY 2 (N=985) | Medtronic Family (N=977)
Pulse generator Related (Cardiac disorders) | 33 (33) | 21 (21)
Right atrial lead related (Cardiac disorders) | 18 (25) | 11 (11)
Right ventricular lead related (Cardiac disorders) | 48 (57) | 60 (77)
Procedure related (Cardiac disorders) | 30 (32) | 25 (26)
Cardiovascular related (Cardiac disorders) | 410 (769) | 373 (690)
Other (Cardiac disorders) | 190 (303) | 174 (239)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No